CLINICAL TRIAL: NCT02991001
Title: The Effect of Hydrodissection for Patients With Carpal Tunnel Syndrome
Brief Title: The Effect of Hydrodissection for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hydrodissection for CTS
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Hydrodissection
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonography; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal saline hydrodissection (Experimental): Ultrasound-guided hydrodissection with normal saline between carpal tunnel and median nerve.
  Interventions: Procedure: Ultrasound-guided hydrodissection; Device: Ultrasound; Drug: Normal Saline
- Normal saline (Placebo Comparator): Ultrasound-guided injection with normal saline at subcutaneous layer beyond the carpal tunnel region
  Interventions: Procedure: Placebo ultrasound-guided injection; Device: Ultrasound; Drug: Normal Saline

INTERVENTIONS:
Procedure: Ultrasound-guided hydrodissection — Ultrasound-guided hydrodissection with 5cc normal saline between carpal tunnel and median nerve.
  Arms: Normal saline hydrodissection
Procedure: Placebo ultrasound-guided injection — Ultrasound-guided injection with 5cc normal saline at subcutaneous layer beyond carpal tunnel
  Arms: Normal saline
Device: Ultrasound
Drug: Normal Saline

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Rather than other progressive disease, CTS is characterized by remission and recurrence. The hydrodissection could decrease the entrapment of nerve to restore blood supply. Despite the hydrodissection was pervasively used in clinical practice, current researches contain small participant without control group or randomized leading to foreseeable selection bias. The investigators design a randomized, double-blind, controlled trail to assess the effect after ultrasound-guided hydrodissection in patients with CTS.

DETAILED DESCRIPTION:
After obtaining written informed consent, patients with bilateral CTS will been randomized into intervention and control group. Participants in intervention group received one-dose ultrasound-guided hydrodissection and control side received one-dose ultrasound-guided injection at subcutaneous layer beyond carpal tunnel. No additional treatment after injection through the study period. The primary outcome is visual analog scale (VAS) and secondary outcomes include Boston Carpal Tunnel Syndrome Questionnaire (BCTQ), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and finger pinch strength. The evaluation was performed pretreatment as well as on the 2nd week, 1st, 2nd and 3rd month after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Cervical radiculopathy
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline of severity of symptoms and functional status on 2nd week, 1st, 2nd, 3rd and 6th month after injection | Pre-treatment, 2nd week, 1st, 2nd and 3rd month after injection
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of CTS which encompasses two components. In total, 11 questions and 8 items were evaluated to rate the symptom severity scale (SSS) and functional status scale (FSS), respectively. Both subscales range from 1 to 5 with a higher score indicating a higher degree of disability. The mean of total SSS and FSS divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 2nd and 3rd month after injection | Pre-treatment, 2nd week, 1st, 2nd , 3rd and 6th month after injection
  Digital pain severity or paresthesia/dysthesia was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain.
Change from baseline of cross-sectional area of the median nerve on 2nd week, 1st, 2nd and 3rd month after injection | Pre-treatment, 2nd week, 1st, 2nd , 3rd and 6th month after injection
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of conduction velocity, amplitude of median nerve on 2nd week, 1st, 2nd and 3rd month after injection | Pre-treatment, 2nd week, 1st, 2nd , 3rd and 6th month after injection
  Antidromic sensory nerve conduction velocity of the median nerve before treatment and multiple time frame after treatment.
Change from baseline of finger pinch on 2nd week, 1st, 2nd and 3rd month after injection | Pre-treatment, 2nd week, 1st, 2nd, 3rd and 6th month after injection
  The finger pinch strength was measured using dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Smith J, Wisniewski SJ, Finnoff JT, Payne JM. Sonographically guided carpal tunnel injections: the ulnar approach. J Ultrasound Med. 2008 Oct;27(10):1485-90. doi: 10.7863/jum.2008.27.10.1485. PMID 18809959
- [Result] DeLea SL, Chavez-Chiang NR, Poole JL, Norton HE, Sibbitt WL Jr, Bankhurst AD. Sonographically guided hydrodissection and corticosteroid injection for scleroderma hand. Clin Rheumatol. 2011 Jun;30(6):805-13. doi: 10.1007/s10067-010-1653-6. Epub 2011 Jan 15. PMID 21234632
- [Result] Choi CK, Lee HS, Kwon JY, Lee WJ. Clinical implications of real-time visualized ultrasound-guided injection for the treatment of ulnar neuropathy at the elbow: a pilot study. Ann Rehabil Med. 2015 Apr;39(2):176-82. doi: 10.5535/arm.2015.39.2.176. Epub 2015 Apr 24. PMID 25932413
- [Result] Chang KV, Hung CY, Ozcakar L. Snapping Thumb and Superficial Radial Nerve Entrapment in De Quervain Disease: Ultrasound Imaging/Guidance Revisited. Pain Med. 2015 Nov;16(11):2214-5. doi: 10.1111/pme.12867. Epub 2015 Jul 27. No abstract available. PMID 26218266
- [Derived] Wu YT, Chen SR, Li TY, Ho TY, Shen YP, Tsai CK, Chen LC. Nerve hydrodissection for carpal tunnel syndrome: A prospective, randomized, double-blind, controlled trial. Muscle Nerve. 2019 Feb;59(2):174-180. doi: 10.1002/mus.26358. Epub 2018 Dec 4. PMID 30339737